CLINICAL TRIAL: NCT03682276
Title: PRIME-HCC: Preliminary Assessment of Safety and Bioactivity of the Ipilimumab and Nivolumab Combination Prior to Liver Resection (LR) in Hepatocellular Carcinoma (HCC)
Brief Title: Safety and Bioactivity of Ipilimumab and Nivolumab Combination Prior to Liver Resection in Hepatocellular Carcinoma
Acronym: PRIME-HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/36/2017; 2018-000987-27 (EudraCT Number); CA209-9LC (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Ipilimumab, solution for infusion, 1 milligram per kilogram body weight, once every 3 weeks, for 3 weeks; Nivolumab, solution for infusion, 3 milligrams per kilogram body weight, once every 3 weeks, for 6 weeks
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: Ipilimumab — Ipilimumab is a monoclonal antibody given as an immunotherapy
  Other Names: YERVOY
Biological: Nivolumab — Nivolumab is a monoclonal antibody given as an immunotherapy
  Other Names: OPDIVO

SUMMARY:
The PRIME-HCC trial will assess the effects of combination treatment with nivolumab (OPDIVO) and ipilimumab (YERVOY) pre-operatively in hepatocellular carcinoma patients for whom liver resection is planned. The trial will be conducted at a small number of National Health Service hospitals in the UK. Participants will receive two doses of nivolumab and a single dose of ipilimumab in the weeks before their planned surgery.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to be conducted in 32 patients at a small number of UK hospitals. The study is in 2 parts: Part 1 will confirm, in a small number of patients, that the treatment regimen is safe and doesn't result in unacceptable delay to liver resection. Part 2 will expand the number of patients studied, and provide the opportunity to assess survival over about 2 years after liver resection. The decision to proceed to Part 2 will be taken with advice from an independent, expert committee.

Patients with early-stage HCC will first undergo screening procedures during a 28-day time window between giving consent and starting drug treatment. Screening procedures will include:

* Medical interview and physical exam
* ECG
* Tumour biopsy
* Tumour imaging by MRI
* Tumour imaging by CT
* Blood and urine samples
* Stool sample (optional)

Patients meeting the protocol-specified criteria will be enrolled and on Day 1 will have the following:

* Medical interview, and physical exam (if required)
* Blood and urine samples
* Intravenous dose of ipilimumab ('YERVOY') 1 milligram per kilogram body weight
* Intravenous dose of nivolumab ('OPDIVO') 3 milligrams per kilogram body weight

On Day 22 the participants will have the following:

* Medical interview, and physical exam (if required)
* Blood and urine samples
* Intravenous dose of nivolumab ('OPDIVO') 3 milligrams per kilogram body weight

On Day 43 the participants will have the following:

* Medical interview, and physical exam (if required)
* ECG
* Tumour imaging by MRI
* Blood and urine samples
* Stool sample (optional)

Patients who remain eligible for liver resection will likely undergo surgery within a few days of the Day 43 visit.

On Day 127 the participants will have the following:

* Medical interview, and physical exam (if required)
* Tumour imaging by MRI
* Blood and urine samples

Every 4 months thereafter until 2 years later, or until starting another anti-cancer treatment, participants will have tumour imaging by MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for the trial.
2. Aged ≥18 years
3. Confirmed diagnosis of HCC
4. Willing to provide tissue from an excisional biopsy of a tumour lesion
5. Have measurable disease by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI) defined by RECIST 1.1 criteria
6. Ineligible for liver transplantation
7. Medically fit to undergo surgery as determined by the treating medical and surgical oncology team
8. ECOG performance status 0 or 1
9. Adequate organ function
10. Overall Child-Pugh class A
11. Female patient of childbearing potential should have a negative serum pregnancy test within 24 h of her first dose of IMP
12. Women of childbearing potential must be willing to use a highly effective method of contraception for the course of the study through 5 months after the last dose of Investigational Medicinal Product (IMP). Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
13. Sexually active males must agree to use an adequate method of contraception starting with the first dose of IMP through 7 months after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

1. Extrahepatic metastasis
2. Prior systemic anticancer treatment for HCC, including an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody
3. Prior orthotopic liver transplantation
4. Any major surgery within the 3 weeks prior to enrolment
5. Hepatic encephalopathy
6. Ascites that is refractory to diuretic therapy
7. Is currently receiving anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy or biologic therapy) or has participated or is participating in a study of an IMP or used an investigational device within 4 weeks of the first dose of IMP
8. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy
9. Known history of active Bacillus Tuberculosis (TB)
10. History of known hypersensitivity to any monoclonal antibody or any of their excipients
11. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
12. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
13. Known history of, or any evidence of active, non-infectious pneumonitis
14. Active infection requiring systemic therapy, with exceptions relating to Hepatitis B and C virus infection
15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Principal Investigator (PI)
16. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
17. Pregnant or breastfeeding
18. Known history of Human Immunodeficiency Virus (HIV; HIV 1/2 antibodies)
19. Received a live vaccine within 30 days of first dose of IMP administration. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Delay to surgery | Up to Day 89
  Number of patients with an unplanned delay to surgery to Day 89 or later
Incidence of treatment-emergent adverse events [Safety and Tolerability] | Up to Day 127
  Safety and tolerability of the nivolumab and ipilimumab combination based on NCI CTCAE v5.0 criteria from the day of first nivolumab and ipilimumab administration to 126 days later

SECONDARY OUTCOMES:
Objective response rate | Up to Day 43
  Objective response rate on pre-resection imaging 42 days after the day of first nivolumab and ipilimumab administration using RECIST v1.1 criteria
Pathologic response rate | Up to Day 88 or up to liver resection, whichever came first
  Pathologic response rate on hematoxylin and eosin evaluation of the resected specimen

CONTACTS AND LOCATIONS:
Overall Officials: David J Pinato, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinato DJ, Cortellini A, Sukumaran A, Cole T, Pai M, Habib N, Spalding D, Sodergren MH, Martinez M, Dhillon T, Tait P, Thomas R, Ward C, Kocher H, Yip V, Slater S, Sharma R. PRIME-HCC: phase Ib study of neoadjuvant ipilimumab and nivolumab prior to liver resection for hepatocellular carcinoma. BMC Cancer. 2021 Mar 23;21(1):301. doi: 10.1186/s12885-021-08033-x. PMID 33757459